CLINICAL TRIAL: NCT04696458
Title: Effects of a Multispecies Probiotic on Migraine: A Randomized Controlled Trial
Brief Title: Effects of a Multispecies Probiotic on Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Health (Other)
Collaborators: Kaneka Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-21-7729
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Migraine; Irritable Bowel Syndrome; Headache, Migraine
Keywords: Probiotics; Headache Disorders; Migraine Disorders; Pain; Digestive System Diseases; Neurologic Manifestations; Gut-Brain Axis; Microbiome; Functional Gastrointestinal Symptoms
MeSH Terms: conditions — Migraine Disorders; Irritable Bowel Syndrome; Headache Disorders; Pain; Digestive System Diseases; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL PROBIOTIC (Experimental): 1 Multistrain Probiotic Capsule
  Interventions: Dietary Supplement: Lactobacillus plantarum (CECT7484 and CECT7485)/ Pediococcus acidilactici (CECT7483)
- Placebo (Placebo Comparator): 1 Identical Placebo Capsule
  Interventions: Other: Placebo Comparator: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum (CECT7484 and CECT7485)/ Pediococcus acidilactici (CECT7483) — Probiotic Capsules in blister packets of capsules containing the probiotic intervention contain a combination of three strains of lactic acid bacteria: two Lactobacillus plantarum (CECT7484 and CECT7485) and one Pediococcus acidilactici (CECT7483).
  Other Names: Placebo Comparator: Placebo
  Arms: EXPERIMENTAL PROBIOTIC
Other: Placebo Comparator: Placebo — Placebo Capsules in blister packets of capsules containing the inert (controlled) non-interventional treatment.
  Other Names: inert placebo
  Arms: Placebo

SUMMARY:
The prevalence of migraine is higher in female patients with various intestinal diseases. An explanation could be that migraine is caused by a leaky gut, defined by increased intestinal permeability that permits particles to pass through the gastrointestinal wall. Probiotics, may be able to improve intestinal barrier function.

OBJECTIVE: To test whether probiotics, as adjucnt therapy, can reduce incidence and severity of migraine attacks by reducing intestinal permeability.

DETAILED DESCRIPTION:
Given the significant unmet need for improved therapies that address migraine disorders and concurrent irritable bowel syndrome (IBS), this study seeks to investigate the impact of probiotics on the sequelae of symptoms associated with both migraine and IBS.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine diagnosis for a minimum of 1 year (12-months)
* Between 3-12 migraine episodes /month
* Comorbid, symptomatic, irritable bowel syndrome during the screening period
* On a steady treatment regimen: preventative and acute migraine medications and therapies unchanged over the last 6 months
* Access to Scripps Center for Integrative Medicine
* Access to smartphone or computer to complete electronic surveys

Exclusion Criteria:

* Other GI or hepatic diagnoses (Inflammatory Bowel Disease (IBD), Small Intestinal Bacterial Overgrowth (SIBO), Non-Alcoholic Fatty Liver Disease (NAFLD), elevated Liver Function Tests (LFTs) within the last 6 months)
* Prior GI surgery
* Prior GI infection in the previous 3-months
* Antibiotic treatment in previous last 3 months
* Diagnosed Autoimmune disease
* Current corticosteroids use
* Morbid obesity (BMI >40)
* Took Probiotics or Probiotic-containing supplements or therapy in the previous 3-months
* Diagnosis of post-traumatic headache or cervicogenic headache
* Pregnancy or plans to become pregnant during study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Migraine-induced Disability as measured by the Migraine Induced Disability Assessment Score (MIDAS) total score | Change day 0 to week 12
  This survey measures headache frequency, disability, severity

SECONDARY OUTCOMES:
Improved Quality of Life (QoL) and reduced depressive symptoms (per Patient Health Questionnaire (PHQ-9)) | Change day 0 to week 12
  Survey used to assess depressive symptoms
Reduced severity of Gastrointestinal (GI) symptoms (per Irritable Bowel Syndrome Severity Scoring System (IBS -SSS)) | Change day 0 to week 12
  Survey used to assess IBS symptoms
Reduced generalized anxiety (per Generalized Anxiety Disorder (GAD-7)) | Change day 0 to week 12
  Survey used to assess anxiety symptoms
Reduce headache parameters (headache episodes, headache days, intensity, duration) based on MIDAS subcomponents and journal/diary | Change day 0 to week 12
  Survey used to assess migraine treatments symptoms
Change in acute medication requirements | Change day 0 to week 12
  Survey used to assess medication requirements

CONTACTS AND LOCATIONS:
Overall Officials: Megan Sweeney, MPH, Study Chair — Scripps Clinic; Kristen Hickey, Study Chair — Scripps Clinic
Locations (1):
- Scripps Center for Integrative Medicine, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data and information can be shared upon request after study completion
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 Months after Study Publication. Can be shared indefinitely
Access Criteria: Email to PI or study director requesting data. Only secure data will be sent via a secure password protected document.

REFERENCES:
- [Background] Arzani M, Jahromi SR, Ghorbani Z, Vahabizad F, Martelletti P, Ghaemi A, Sacco S, Togha M; School of Advanced Studies of the European Headache Federation (EHF-SAS). Gut-brain Axis and migraine headache: a comprehensive review. J Headache Pain. 2020 Feb 13;21(1):15. doi: 10.1186/s10194-020-1078-9. PMID 32054443
- [Background] Dai YJ, Wang HY, Wang XJ, Kaye AD, Sun YH. Potential Beneficial Effects of Probiotics on Human Migraine Headache: A Literature Review. Pain Physician. 2017 Feb;20(2):E251-E255. PMID 28158162
- [Background] Loren V, Manye J, Fuentes MC, Cabre E, Ojanguren I, Espadaler J. Comparative Effect of the I3.1 Probiotic Formula in Two Animal Models of Colitis. Probiotics Antimicrob Proteins. 2017 Mar;9(1):71-80. doi: 10.1007/s12602-016-9239-5. PMID 27832441
- [Background] Lorenzo-Zuniga V, Llop E, Suarez C, Alvarez B, Abreu L, Espadaler J, Serra J. I.31, a new combination of probiotics, improves irritable bowel syndrome-related quality of life. World J Gastroenterol. 2014 Jul 14;20(26):8709-16. doi: 10.3748/wjg.v20.i26.8709. PMID 25024629
- [Background] Naghibi MM, Day R, Stone S, Harper A. Probiotics for the Prophylaxis of Migraine: A Systematic Review of Randomized Placebo Controlled Trials. J Clin Med. 2019 Sep 11;8(9):1441. doi: 10.3390/jcm8091441. PMID 31514352
- [Background] National Institute of Neurological Disorders and Stroke. Headache: Hope Through Research. April 2016.